CLINICAL TRIAL: NCT04485962
Title: Treatment of Patients With Skin Burns Using Autologous Keratinocytes and Skin Fibroblasts
Brief Title: Treatment of Patients With Skin Burns Using Keratinocytes and Skin Fibroblasts
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian Medical Academy of Post-Graduate Education (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_Fibr(Burns)
Record Dates: First submitted 2020-07-17; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Burns
Keywords: burns; fibroblasts; keratinocytes
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fibroblasts and keratinocytes treated patients (Experimental): Fibroblasts and keratinocytes treated patients
  Interventions: Biological: Fibroblasts and keratinocytes

INTERVENTIONS:
Biological: Fibroblasts and keratinocytes — Autologous cultured fibroblasts and keratinocytes
  For PR: The name " fibroblasts and keratinocytes" is exactly the name of the cell product registered by our ministry of health. There is no trade or international name.

SUMMARY:
Treatment of patients with burns of the skin of the 2nd degree using: autologous keratinocytes and skin fibroblasts mixed with collagen gel 7% (tissue equivalent of the skin)

DETAILED DESCRIPTION:
Treatment of patients with burns of the skin of the 2nd degree by applying a wound covering with layer-by-layer cultured autologous keratinocytes and fibroblasts in collagen gel

ELIGIBILITY:
Inclusion Criteria:

* skin burns of the 2nd degree

Exclusion Criteria:

* acute and chronic infectious diseases: HIV, viral hepatitis, tuberculosis
* mental disorders
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of cured patients | 1 month
  Number of patients cured
Number of patients with treatment-related adverse events | 1 month
  Cell application related adverse events assessed by blood count, liver and function tests

CONTACTS AND LOCATIONS:
Overall Officials: Igor Volotovski, Prof, Study Director — Head of the Lab of Institute of Biophysics and Cell Engineering; Vladimir Podgaiskiy, Prof, Study Director — Head of the plastic surgery and combustiology; Alexey Chasnoit, Dr, Principal Investigator — Dean of the plastic surgery and combustiology; Zinaida Kvacheva, Dr, Principal Investigator — Lead Researcher of Institute of Biophysics and Cell Engineering
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No